CLINICAL TRIAL: NCT03847519
Title: A Phase 1/2, Open-Label Study of ADXS-503 Alone and in Combination With Pembrolizumab in Subjects With Metastatic Squamous or Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Study of ADXS-503 With or Without Pembro in Subjects With Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advaxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADXS-503-101
Record Dates: First submitted 2019-01-08; First posted 2019-02-20 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer, Non-Small Cell; Metastatic Squamous Cell Carcinoma; Metastatic Non-Squamous Cell Carcinoma
Keywords: NSCLC Lung Cancer; Metastatic Squamous Non-Small Cell Lung Cancer; Metastatic Non-Squamous Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell | interventions — A 503; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Safety phase:
  * Part A: ADXS-503 monotherapy dose escalation
  * Part B: ADXS-503 + pembrolizumab dose escalation
  Efficacy phase:
  • Part C: ADXS-503 + pembrolizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Phase Part A (Experimental): Enroll subjects with metastatic squamous or non-squamous NSCLC who have become refractory or intolerant to standard therapy. ADXS-503 monotherapy will be evaluated at 2 planned escalating dose levels:
  * Dose level 1: 1e8 CFU of ADXS-503, IV, every 3 weeks until disease progression, unacceptable toxicity, or another treatment discontinuation criterion is met.
  * Dose level 2: 5e8 CFU of ADXS-503, IV, every 3 weeks until disease progression, unacceptable toxicity, or another treatment discontinuation criterion is met.
  Interventions: Drug: ADXS-503
- Safety Phase Part B (Experimental): Enroll subjects with metastatic squamous or non-squamous NSCLC. ADXS-503 will be evaluated at 2 planned escalating dose levels in combination with a fixed dose of pembrolizumab:
  * Dose level 1: 1e8 CFU of ADXS-503 + 200 mg of pembrolizumab, IV, every 3 weeks for up to 2 years or until disease progression, unacceptable toxicity, or another treatment discontinuation criterion is met.
  * Dose level 2: 5e8 CFU of ADXS-503 + 200 mg of pembrolizumab, IV, every 3 weeks for up to 2 years or until disease progression, unacceptable toxicity, or another treatment discontinuation criterion is met. (recruitment is on hold for this arm)
  Interventions: Drug: ADXS-503; Drug: Pembrolizumab
- Efficacy Phase Part C (Experimental): Enroll subjects with metastatic squamous or non-squamous NSCLC.
  1e8 CFU of ADXS-503 + 200 mg of pembrolizumab, IV, every 3 weeks for up to 2 years or until disease progression, unacceptable toxicity, or another treatment discontinuation criterion is met.
  Interventions: Drug: ADXS-503; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ADXS-503 — A live attenuated Listeria monocytogenes (Lm)-based immunotherapy bioengineered to elicit T cell responses against shared tumor antigens commonly found in patients with squamous and non-squamous NSCLC.
  Other Names: Lm immunotherapy; A503
Drug: Pembrolizumab — a programmed death receptor-1 (PD-1)- blocking antibody.
  Other Names: Keytruda; pembro
  Arms: Efficacy Phase Part C; Safety Phase Part B

SUMMARY:
A Phase 1/2, Open-Label Study of ADXS-503 Alone and in Combination with Pembrolizumab in Subjects with Metastatic Squamous or Non-Squamous Non-Small Cell Lung Cancer

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of ADXS-503, administered as monotherapy in Part A and in combination with pembrolizumab in Part B, and to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD). As well, to characterize the preliminary anti-tumor activity of ADXS-503, administered in combination with pembrolizumab in Part C, per RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Subject and/or their legally authorized representative must be capable of understanding the investigational nature, potential risks, and benefits of the study. The subject and/or their legally authorized representative must sign a written informed consent;
2. Subject is ≥18 years of age upon signing the Informed Consent Form;
3. Subject has histologically or cytologically confirmed stage IV (metastatic) squamous or non-squamous NSCLC

   * Part A only:

     ▪ Subject has received, and then progressed or been intolerant to up to 3 lines of prior therapy in the metastatic setting, including approved chemotherapy, targeted therapy, immunotherapy and antibody therapy, if eligible. Subjects who have received >3 lines of prior therapy may be eligible for Part A, upon discussion with and approval by the Sponsor.
     * Subjects will be eligible for Part A irrespective of PD-L1 expression.
     * Subjects will be eligible for Part A irrespective of EGFR or ALK mutation status. However, subjects with an EGFR sensitizing mutation or ALK translocation must have received and then progressed or been intolerant to at least 1 prior line of approved targeted therapy to be eligible for Part A.
   * Part B only:

     * Subject is undergoing treatment with pembrolizumab monotherapy for metastatic NSCLC
     * Subject's most recent tumor assessment is consistent with PD according to RECIST v1.1
     * The Investigator has determined that PD should be confirmed within 4-8 weeks, and pembrolizumab treatment will continue pending PD confirmation
     * Subject is willing to undergo a confirmatory scan 4-8 weeks from the prior scan that indicated progression on pembrolizumab
     * There is no evidence of rapid disease progression or clinical deterioration in the subject that would preclude continuation of pembrolizumab treatment pending confirmation of PD.
   * Part C only:

     * Subject has received no prior systemic treatment in the metastatic setting. Subjects previously treated with adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months prior to the diagnosis of metastatic disease.
     * Subject has provided a formalin-fixed tumor sample from a biopsy of a tumor lesion either at the time of or after the diagnosis of metastatic disease AND from a site not previously irradiated, to assess for PD-L1 status. Biopsies obtained PRIOR to the administration of any systemic therapy to treat the subject's tumor (such as neoadjuvant/adjuvant therapy) will not be permitted for analysis. The tissue sample must be received by the central laboratory vendor prior to enrollment. Fine needle aspirates, Endobronchial Ultrasound (EBUS) or cell blocks are not acceptable. Needle or excisional biopsies, or resected tissue is required. If the tumor specimen is not evaluable for PD-L1 expression by the central laboratory, an additional tumor specimen may be submitted.
     * Subject's tumor has PD-L1 expression of ≥50%, as determined by immunohistochemistry (IHC) at a central laboratory.
     * Subject's tumor does not harbour an EGFR sensitizing (activating) mutation or ALK translocation. EGFR sensitizing mutations are mutations that are amenable to treatment with TKIs (e.g., erlotinib, gefitinib, afatanib, osimertinib). ALK translocations are amendable to treatment with TKIs such as crizotinib, alectinib and ceritinib. Investigators must produce the source documentation of the EGFR mutation and ALK translocation status in all subjects with non-squamous histology AND for subjects in whom testing is clinically indicated. If either an EGFR sensitizing mutation or ALK translocation is detected, additional information regarding the mutation status of the other molecule is not required. If the clinical site is unable to provide the source documentation, EGFR and ALK testing should be performed per institutional standard of care.
4. Subject has measurable disease for response assessment as defined by RECIST v1.1 by the Investigator;
5. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 (see Appendix 11);
6. Subject has a life expectancy of at least 3 months;
7. Subject has recovered to Grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.03 (NCI-CTCAE v4.03) of all clinically significant toxic effects of prior anti-cancer chemotherapy, immunotherapy, radiotherapy or surgery before entering this study, except for alopecia;
8. Subject has no major existing comorbidities or medical conditions that would preclude therapy in the opinion of the Investigator;
9. Subject has adequate organ function
10. A female subject is eligible to participate if she is not pregnant (see Appendix 5), not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 5 OR
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 5 during the treatment period and for at least 120 days after the final dose of study treatment;
11. A female subject of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study treatment and throughout the study as defined in the SoA. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. A male subject is eligible if he agrees to follow the contraceptive guidance in Appendix 5 during the treatment period and for at least 120 days after the final dose of study treatment.

Exclusion Criteria:

1. Subject has an ongoing different primary malignancy. Exceptions include treated basal cell carcinoma of the skin or squamous cell carcinoma of the skin;
2. Subject has an active autoimmune disease requiring systemic treatment within the past 3 months, a documented history of clinically severe autoimmune disease, or a disorder that requires systemic corticosteroids or immunosuppressive agents. Subjects with vitiligo, psoriasis, alopecia or resolved childhood asthma/atopy not requiring systemic treatment would be an exception to this rule. Subjects with hypothyroidism who are stable on hormone replacement (>10 mg daily prednisone equivalent) or Sjögren's syndrome will not be excluded from the study;
3. Subject has a diagnosis of primary immunodeficiency, is dependent on or has received systemic corticosteroid therapy (>10 mg daily prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study treatment. Inhaled or topical corticosteroids, and adrenal replacement corticosteroid doses >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease;
4. Subject has neuropathy (sensory or motor) ≥Grade 3 per CTCAE v4.03;
5. Subject has had an allogeneic tissue/solid organ transplant;
6. Subject has interstitial lung disease (ILD) OR has had a history of pneumonitis that has required oral or IV steroids;
7. Subject has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (no new or enlarging brain metastases) by imaging for at least 2 weeks following treatment, and clinically stable with no symptoms due to CNS metastasis, and are not using corticosteroids for at least 14 days prior to the start of study treatment;
8. Subject has a concurrent unstable or uncontrolled medical condition (e.g., active uncontrolled systemic infection, unstable angina, congestive heart failure, uncontrolled diabetes) or other chronic disease, which in the opinion of the Investigator could compromise the subject or the study;
9. Subject has a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies);
10. Subject has a known active hepatitis B (e.g., HBsAg reactive) or hepatitis C infection (e.g., HCV RNA [qualitative] is detected) or tuberculosis;
11. Subject has an active infection requiring systemic therapy or is dependent on or currently receiving antibiotics that cannot be discontinued before dosing. (Note: Subjects who discontinue an antibiotic prior to dosing must wait at least 5 half-lives after the last dose of antibiotic before receiving any study treatment);
12. Subject has known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the study;
13. Subject has an implanted medical device that poses a high risk for bacterial colonization and/or that cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screws, metal plates, bone grafts, or other exogenous implants). NOTE: More common devices and prosthetics that include arterial and venous stents, dental and breast implants and venous access devices (e.g., Port-a-Cath or Mediport) are permitted. Sponsor must be contacted prior to consenting any subject who has any other device or implant;
14. Subject is pregnant or breastfeeding, or plans to become pregnant or to father children, from the Screening visit through at least 120 days after the final dose of study treatment;
15. Subject has a contraindication (e.g., sensitivity/allergy) to trimethoprim/ sulfamethoxazole and ampicillin;
16. Subject has a contraindication to non-steroidal anti-inflammatory drugs (NSAIDs);
17. Subject has a known allergy to any component of the study formulation(s);
18. Subject has a history of listeriosis;
19. Subject has any other serious or uncontrolled physical or mental condition/disease that, as judged by the Investigator, could place the subject at higher risk derived from their participation in the study, could confound results of the study, or would be likely to prevent compliance with the requirements of the study;
20. Subject has received chemotherapy and/or radiation therapy (except palliative radiation therapy for disease-related pain) within 2 weeks of the first dose of study treatment;
21. Subject has received monoclonal antibody or other biologic therapy within 5 half-lives or 28 days prior to the first dose of study treatment, whichever is shorter. An exception to this exclusion criterion will be pembrolizumab monotherapy for subjects enrolled in Part B;
22. Subject has received prior treatment with an Lm-based immunotherapy;
23. Subject is receiving or plans to receive future treatment with PI3K or TNFα inhibitors;
24. Subject has received a live vaccine within 30 days prior to the first dose of study treatment;
25. Subject has not recovered to baseline from AEs, with the exception of alopecia, due to previously administered agent(s);
26. Subject has had major surgery within 6 weeks prior to the initiation of study treatment. NOTE:

    All surgical complications must have recovered to baseline or Grade ≤1 prior to the initiation of study therapy. Sponsor must be consulted prior to enrolling subjects on the study who recently had a major surgery or have a new artificial implant, and/or devices;
27. Subject is currently participating in or has participated in a study of an investigational agent(s) within 4 weeks of the first dose of study treatment;
28. Subject is or has an immediate family member (spouse or children) who, as investigational site or sponsor staff, is directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific subject;

    Exclusion Criteria for Part C only
29. In Part C, subject has received systemic therapy for the treatment of their metastatic NSCLC.

    Completion of treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease;
30. In Part C, subject has an EGFR sensitizing mutation and/or an ALK translocation;
31. In Part C, baseline tumor specimen is not evaluable for PD-L1 expression by the central laboratory. If an additional tumor specimen is submitted AND evaluable for PD-L1 expression, the subject will be eligible to participate if PD-L1 expression is assessed as ≥50% by the central laboratory;
32. In Part C, subject has received prior systemic chemotherapy, biological therapy, OR major surgery within 6 weeks of the first dose of study treatment; received thoracic radiation therapy of >30 Gy within 6 months of first dose of study treatment;
33. In Part C, subject has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti- CD137, or anti-CTLA-4 antibody, or any other antibody or drug that specifically targets T cell co-stimulation or immune checkpoint pathways.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Surya Vangala, Study Director — Senior Director, Clinical Operations, Advaxis Inc
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Illinois CancerCare, P.C., Peoria, Illinois
  - The University of Kansas Medical Center, Westwood, Kansas
  - Atlantic Health System, Carol G Simon Cancer Center, Morristown, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Providence Cancer Institute, Portland, Oregon
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A Phase 1/2, Open-Label Study of ADXS-503 Alone and in Combination with Pembrolizumab in Subjects with Metastatic Squamous or Non-Squamous Non-Small Cell Lung Cancer. Protocol ADXS-503-101, Advaxis Inc, 2018.

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Phase Part A - ADXS-503: 1e8 CFU of ADXS-503, IV, every 3 weeks until disease progression, unacceptable toxicity, or another treatment discontinuation criterion is met.
- Safety Phase Part B - ADXS-503 + 200mg Pembrolizumab: 5e8 CFU of ADXS-503 + 200 mg of pembrolizumab, IV, every 3 weeks for up to 2 years or until disease progression, unacceptable toxicity, or another treatment discontinuation criterion is met.
- Efficacy Phase Part C - ADXS-503 + 200mg Pembrolizumab: 1e8 CFU of ADXS-503 + 200 mg of pembrolizumab, IV, every 3 weeks for up to 2 years or until disease progression, unacceptable toxicity, or another treatment discontinuation criterion is met.
Period: Overall Study
Arm/Group | Safety Phase Part A - ADXS-503 | Safety Phase Part B - ADXS-503 + 200mg Pembrolizumab | Efficacy Phase Part C - ADXS-503 + 200mg Pembrolizumab
Started | 7 | 14 | 3
Completed | 1 | 1 | 0
Not Completed | 6 | 13 | 3
Not completed — Death | 5 | 8 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Study Terminated by Sponsor | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: All Treated Subjects Population includes subjects enrolled in the study who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Phase Part A - ADXS-503 | Safety Phase Part B - ADXS-503 + 200mg Pembrolizumab | Efficacy Phase Part C - ADXS-503 + 200mg Pembrolizumab | Total
Number analyzed (Participants) | 7 | 14 | 3 | 24
Age, Continuous [Mean (Full Range); unit: years] | 65.7 [56 to 83] | 68.3 [55 to 87] | 70.7 [68 to 75] | 68.2 [55 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 1 | 12
  Male | 3 | 7 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 7 | 10 | 2 | 19
  Unknown or Not Reported | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety/Tolerability of ADXS-503 Monotherapy in Part A and ADXS-503 With Pembrolizumab in Part B: Graded Per Comment Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: The safety/tolerability of ADXS-503 monotherapy in Part A and in combination pembrolizumab in Part B was assessed by the number of patients with treatment-related adverse events.
Time Frame: 12 Months
Population: All Treated Subjects Population will include subjects enrolled in the study arms A and B who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Phase Part A - ADXS-503 | Safety Phase Part B - ADXS-503 + 200mg Pembrolizumab
Number analyzed (Participants) | 7 | 14
Participants | 4 | 11

2. Primary Outcome: Preliminary Anti-tumor Activity of ADXS-503 + Pembrolizumab in Part C as Assessed by the Objective Response Rate (ORR)
Description: The anti-tumor activity of ADXS-503 + pembrolizumab was assessed by the objective response rate (ORR). The ORR according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 was defined as the number of participants with objective evidence of radiologic complete response (CR: the disappearance of all target lesions) and partial response (PR: at least 30% decrease in the sum of the longest diameters of target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions) as determined from investigator response assessments. Disease Control Rates are based upon confirmed events only.
Time Frame: 3 years
Population: All Treated Subjects Population will include subjects enrolled in Part C of the study who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Efficacy Phase Part C - ADXS-503 + 200mg Pembrolizumab
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Preliminary Anti-tumor Activity of ADXS-503 Alone in Part A and ADXS-503 With Pembrolizumab in Part B as Assessed by the Objective Response Rate (ORR)
Description: The anti-tumor activity of ADXS-503 as monotherapy or in combination with pembrolizumab was assessed by the objective response rate (ORR). The ORR according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 was defined as the number of participants with objective evidence of radiologic complete response (CR: the disappearance of all target lesions) and partial response (PR: at least 30% decrease in the sum of the longest diameters of target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions) as determined from investigator response assessments. Disease Control Rates are based upon confirmed events only.
Time Frame: 3 years
Population: All Treated Subjects Population will include subjects enrolled in Part A and B of the study who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Phase Part A - ADXS-503 | Safety Phase Part B - ADXS-503 + 200mg Pembrolizumab
Number analyzed (Participants) | 7 | 13
Participants | 0 | 1

4. Secondary Outcome: Safety/Tolerability of ADXS-503 With Pembrolizumab in Part C: Graded Per Comment Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: The safety/tolerability of ADXS-503 in combination with pembrolizumab in Part C was assessed by the number of patients with treatment-related adverse events.
Time Frame: 3 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Efficacy Phase Part C - ADXS-503 + 200mg Pembrolizumab
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: 3 years
Description: All Treated Subjects Population include subjects enrolled in the study who received at least one dose of study medication
Arm/Group | Safety Phase Part A - ADXS-503 | Safety Phase Part B - ADXS-503 + 200mg Pembrolizumab | Efficacy Phase Part C - ADXS-503 + 200mg Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 5/7 | 8/14 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/14 | 3/3
Other Adverse Events (participants affected / at risk) | 7/7 | 13/14 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Phase Part A - ADXS-503 (N=7) | Safety Phase Part B - ADXS-503 + 200mg Pembrolizumab (N=14) | Efficacy Phase Part C - ADXS-503 + 200mg Pembrolizumab (N=3)
Cardiac aneurysm (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Generalized anxiety disorder (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Phase Part A - ADXS-503 (N=7) | Safety Phase Part B - ADXS-503 + 200mg Pembrolizumab (N=14) | Efficacy Phase Part C - ADXS-503 + 200mg Pembrolizumab (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 5 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 2
Chills (General disorders) | 1 | 5 | 1
Extravasation (General disorders) | 0 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 6 | 2
Influenza like illness (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 3 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 7 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Ear infection fungal (Infections and infestations) | 0 | 1 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT03847519/Prot_SAP_000.pdf